CLINICAL TRIAL: NCT04368780
Title: The Effect Of Progressive Relaxation Exercises On The Care Satisfaction, Caregiver Burden and The Level of Depression Among Caregivers of Bedridden Elderly Patients
Brief Title: The Effect Of Progressive Relaxation Exercises On The Care Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Sadet ÇAPACI, 2019/24, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/24
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Caregiver
Keywords: caregiver; older people; depression; progressive muscle relaxation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: No Intervention: Control group Experimental: Experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Individuals who provide home care to an elderly person who is dependent on the bed
- Experimental group (Experimental): Individuals who provide home care to an elderly person who is dependent on the bed. It is planned that the exercises will be conducted two days a week with the researcher and on the other days by the caregiver herself for a total of eight weeks.
  Interventions: Other: Effect of Progressive Muscle Relaxation Combined With Music

INTERVENTIONS:
Other: Effect of Progressive Muscle Relaxation Combined With Music — The CD on relaxation exercises developed by the Turkish Psy-chological Associationwas used.In the second of CD 30-min section; relaxation exercises are explained to the accompaniment ofrunning water sounds and verbal instructions. Progressive relaxation technique includes stretching and relaxing the bigmuscle groups (hands, arms, neck, shoulders, face, chest, abdomen,hip, feet andfingers) in the human body on purpose. When steps ofProgressive Relaxation Exercises are analyzed, it is observed thatlearning how to take correct and deep breaths is the most impor-tant step towards learning relaxation. In addition, taking correct breaths is used as a part of the exercise among all relaxation exercises.Steps of Progressive Relaxation Exercise:- breathing exercises- lower extremity exercises- upper extremity exercises- exercise of respiratory muscles.
  Arms: Experimental group

SUMMARY:
The increase in the elderly population, insufficiencies in chronic diseases cause an increase in the number of dependent and dependent elderly. This situation negatively affects caregivers with elderly individuals. nonpharmacological interventions are commonly used to reduce the negative emotions of caregivers due to care. One of these applications is progressive relaxation exercises. This study was planned in a randomized controlled experimental study design to investigate the effect of progressive muscle relaxation exercise. on care satisfaction, care burden and depression level of caregivers who care for bed dependent elderly individuals. The study will consist of 10 interventions, 10 control groups, and 20 caregivers.

DETAILED DESCRIPTION:
Today, changes and developments in technology and lifestyles have lengthened average life span and increased the elderly population. The physical and cognitive changes, health problems, new roles such as being retired or widowed and economic losses come one after another for the elderly, and this turns the old age into a period full of difficul ties. Due to these changes in individuals with aging, older individuals make dependent and dependent on care. Caregivers experience care burdens, emotional stress, depression and anxiety during the care process. There are various non-pharmacological applications in the literature aimed at reducing the level of depression and care burden of caregivers. The non-pharmacological methods used in this study for older people's included progressive muscle relaxation exercise.

Objective: In this study, it is aimed to determine the effect of progressive muscle relaxation exercise. on care satisfaction, care burden and depression level of caregivers of bedridden elderly individuals.

Methodology: This is randomized clinical test. The study will consist of 10 interventions, 10 control groups, and 20 caregivers. The progressive muscle relaxation technique combined with music was employed. In order to collect the data, we adopted the interview with form filling technique, using the introductory information form, The Carer's Assessment Of Satısfactıon Index (Cası-TR), the Zarit Caregiver Burden Scale (ZCBS); and the Beck Depression Scale (BDS).

ELIGIBILITY:
Inclusion Criteria:

* The age of the caregiver is 18 years old.
* Giving care to the elderly patient who is dependent on the bed for at least 3 months and above,
* No psychiatric disease diagnosed,
* No vision, speech or hearing problems that would prevent the information given from being understood and the implementation of PMR exercise,
* Individuals providing voluntary care will be included in participating in the research.

Exclusion Criteria:

* The age of the caregiver under 18
* Giving care to an elderly person dependent on bed for less than 3 months
* With a diagnosis of psychiatric illness
* Has a vision, speech or hearing problem that will prevent the information given from being understood and the implementation of the PMR exercise,
* Caregivers who do not agree to participate in the research will not be included in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
the Carer's Assessment of Satisfaction Index | 2 months
  The caregivers measure satisfaction with care.

SECONDARY OUTCOMES:
the Zarit Caregiver Burden Scale | 2 months
  Assesses the burden of caregivers.
the Beck Depression Scale | 2 months
  Assesses the level of depression of caregivers.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Aksaray University Faculty of Health Science, Aksaray
  - Aksaray University Health Science Faculty, Aksaray

IPD SHARING:
Plan to Share IPD: No
We have no plans.